CLINICAL TRIAL: NCT00469976
Title: Phase II Trial of Enzastaurin Plus Carboplatin and Gemcitabine (ECoG) in Bevacizumab-Ineligible Patients and Enzastaurin Plus Carboplatin, Gemcitabine and Bevacizumab (B-ECoG) in Bevacizumab-Eligible Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Enzastaurin, Carboplatin, and Gemcitabine With or Without Bevacizumab in Treating Patients With Recurrent, Stage IIIB, or Stage IV Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: ECOG will not proceed with activation
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000542546; ECOG-E3506
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bevacizumab
Drug: carboplatin
Drug: enzastaurin hydrochloride
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Enzastaurin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as carboplatin and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving enzastaurin together with carboplatin and gemcitabine, with or without bevacizumab, may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving enzastaurin together with carboplatin and gemcitabine, with or without bevacizumab, works in treating patients with recurrent, stage IIIB, or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the progression-free survival in patients with recurrent or stage IIIB or IV non-small cell lung cancer treated with carboplatin, gemcitabine, and enzastaurin with or without bevacizumab.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the overall survival in patients treated with this regimen.
* Determine the response rate in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 2 treatment groups based on eligibility for bevacizumab therapy.

* Group 1 (bevacizumab-eligible): Patients receive carboplatin IV over 30 minutes and bevacizumab IV over 30-90 minutes on day 1; gemcitabine hydrochloride IV over 30 minutes on days 1 and 8; and oral enzastaurin hydrochloride 3 or 4 times daily on days 1-21 in courses 1-6 and bevacizumab IV over 30-90 minutes on day 1 and oral enzastaurin hydrochloride 3 times daily on days 1-21 in all subsequent courses.
* Group 2 (bevacizumab-ineligible): Patients receive carboplatin, gemcitabine hydrochloride, and enzastaurin hydrochloride as in group 1 in courses 1-6 and enzastaurin hydrochloride alone 3 times daily on days 1-21 in all subsequent courses.

In both groups, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for up to 5 years.

PROJECTED ACCRUAL: A total of 99 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIB (with confirmed malignant pleural effusion), stage IV, or recurrent disease
  * Mixed tumors categorized by the predominant cell type are allowed provided no small cell elements exist

    * Cytologic or histologic elements can be established on metastatic tumor aspirates or biopsy
* Measurable disease as defined by RECIST criteria
* No squamous cell carcinoma (group 1)
* No history of brain metastases (group 1)

  * History of treated brain metastases allowed provided patient is not taking steroids and anti-seizure mediation (group 2)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 mg/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN (≤ 5 times ULN with liver metastases)
* AST and ALT ≤ 3 times ULN (≤ 5 times ULN with liver metastases)
* INR < 1.5 or PTT normal (group 1)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during (groups 1 and 2) and for 6 months after completion of study treatment (group 1)
* No preexisting peripheral neuropathy ≥ grade 2
* Must be able to swallow tablets
* No cardiovascular condition, including any of the following:

  * Myocardial infarction within the past 6 months
  * Cerebrovascular ischemia or stroke within the past 6 months
  * NYHA congestive heart failure > class II
  * Unstable angina pectoris
  * Serious cardiac arrhythmia requiring medication
  * Significant vascular disease
  * Symptomatic peripheral vascular disease
* No concurrent medical condition, psychiatric illness, or limitations that would limit study compliance
* No ongoing active infection or ongoing fever within the past 6 months
* No history of uncontrolled hypertension, defined as blood pressure ≥ 150/90 mm Hg despite being on a stable regimen of anti-hypertensive therapy
* No serious nonhealing wound, ulcer, or bone fracture within the past 4 weeks
* No ongoing or active infection
* No history of thrombotic or hemorrhagic disorders, bleeding diathesis, or coagulopathy (group 1)
* No bleeding > grade 2 or any bleeding requiring intervention within the past 4 weeks (group 1)
* No history of gross hemoptysis (defined as > ½ teaspoon of bright red blood) (group 1)
* Urine protein:creatinine (UPC) ratio < 1.0 by spot urinalysis

  * For UPC ratio > 0.5, a 24-hour urine protein must be obtained and the urine protein level must be < 1,000 mg (group 1)
* None of the following conditions (group 1):

  * Grade II or greater peripheral vascular disease
  * Abdominal fistula
  * Gastrointestinal perforation
  * Intra-abdominal abscess
* No known hypersensitivity to any component of bevacizumab (group 1)
* No history of hypertensive crisis or hypertensive encephalopathy (group 1)

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior major surgical procedure
* More than 7 days since prior minor surgical procedure
* No prior chemotherapy for advanced NSCLC

  * Postoperative adjuvant chemotherapy for previously resected NSCLC allowed if last dose was given > 1 year ago
* More than 3 weeks since prior radiation therapy and recovered
* More than 3 weeks since prior immunotherapy and/or hormonal therapy (not including hormone replacement therapy or contraceptives) and recovered
* More than 14 days since prior enzyme inducing anti-epileptic drugs (EIAEDs)
* More than 10 days since prior and no concurrent daily treatment with acetylsalicylic acid (> 325 mg/day) or NSAIDs known to inhibit platelet function for chronic conditions (group 1)
* No concurrent major surgical procedure (group 1)
* No concurrent carbamazepine, phenobarbital, or phenytoin
* No concurrent therapeutic anticoagulation (group 1)

  * Prophylactic anticoagulation of venous access devices is allowed
* No concurrent treatment with dipyridamole, ticlopidine, clopidogrel, or cilostazol (group 1)
* No concurrent combination antiretroviral therapy for HIV-positive patients

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06

PRIMARY OUTCOMES:
Progression-free survival at 6 months (group 1)
Progression-free survival at 4.5 months (group 2)

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Argiris, MD, Study Chair — University of Pittsburgh; Chandra P. Belani, MD — Milton S. Hershey Medical Center